CLINICAL TRIAL: NCT05280639
Title: Ankle and Pilon Fracture Post Operative Rehabilitation: A Randomized Control Trial Exploring a Simplified Wooden Block Protocol
Brief Title: Simplified Post Op Rehabilitation for Ankle and Pilon Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Seth Yarboro, MD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR200191
Record Dates: First submitted 2021-09-28; First posted 2022-03-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Ankle Fractures; Pilon Fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simplified block protocol (Experimental): subjects in this group will perform a simplified post operative rehabilitation program using a simplified wooden block protocol
  Interventions: Device: Wooden block
- Usual care (Active Comparator): Subjects in this group will perform formal physical therapy or a home exercise program consistent with AAOS standards.
  Interventions: Other: Formal physical therapy or Home Exercise Program

INTERVENTIONS:
Device: Wooden block — Individuals randomized to this group will be given a wooden block at no cost to them and a simplified version of home, self-guided exercises with instructions on how to do the exercises and how often to do so.
  Arms: Simplified block protocol
Other: Formal physical therapy or Home Exercise Program — Individuals randomized to this group will receive the standard formal physical therapy which are sessions run by a physical therapist, usually 2-3 times a week to rehabilitate their ankle OR follow a standardized home exercise program which will be done by yourself with exercise outlined with how they should be performed and how often
  Arms: Usual care

SUMMARY:
The aim of this study is to compare standard post operative rehabilitation with a simplified wooden block stretching protocol that will yield similar results.

DETAILED DESCRIPTION:
Ankle fractures and pilon fractures represent common injuries in orthopedics. These injuries are addressed with re-aligning the bones with surgery, and in some particular cases, they are treated closed reduction and immobilization during healing. The trauma to the ankle as a result of the injury, the prolonged immobilization in a cast or splint and the scar tissue formed during surgery often lead to post injury and post-operative stiffness. Many patients have limited ability to flex the ankle upward (dorsiflexion) following cast or splint removal for these injuries. Physical therapy and rehabilitation represent an an industry-accepted practice for alleviating stiffness and improving function. Currently there are varying studies on the benefits of manual therapy or passive stretch when compared with exercise alone. Neither a supervised exercise program such as formal physical therapy nor a home exercise regiment offer a clear benefit over the other, leading to the question of, if this process can be further simplified to use with the wooden block.

The main functional complaint of patients is "stiffness" or decreased range of motion is in dorsiflexion of the ankle and is cited at approximately 77% of patients following cast or splint removal. This motion is key when walking normally, descending stairs or kneeling and is important to a greater degree when walking up hills , running or rising from a chair. These activities require 10 degrees passive dorsiflexion and 20 degrees on average, respectively. The functional effects of limited ankle dorsiflexion sometimes results in the need for a shoe heel insert or additional surgical procedures to free up the scar in the front of the ankle.

This randomized control trial aims to analyze two currently-used standards of care for ankle and tibial plafond injuries, simplifying the standard post-operative physical therapy/rehabilitation regiment, which would begin a the time of rigid splint removal, when stretching and range of motion is tolerated. Weight bearing with ambulation is slowly adjusted for the weeks following this. This simplified wooden block protocol ankle exercises focus strictly on ankle dorsiflexion using a wooden block. The investigators aim of doing so is to increase compliance with the exercises and with an improved functional outcome as compared with the standard, more complex exercises and time burdensome options.

The aim of this study is to compare the standard post injury/surgery rehabilitation with this new simplified wooden block stretching protocol and analyze the simplified protocol's effectiveness verses other industry accepted exercises/therapy regiments. This study will evaluate pain scores, compliance, range of motion of the ankle and include a Lower Extremity Functionality Score survey, over the course of 3 standard post-operative visits following the subjects injury.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Surgically treated open or closed fractures of the ankle or tibial plafond

Exclusion Criteria:

* Contralateral lower extremity injuries that would limit weight bearing after 6 weeks
* Severe injury requiring flap coverage or vascular reconstruction (Gustilo-Anderson Type IIIB and C respectively)
* Neurological deficits that would impede ability to stand safely unassisted for home exercise regiment
* Desire to participate in formal physical therapy program
* Additional injury that would compromise subjects ability to follow either Home Exercise Program
* Non ambulatory prior to injury
* Previous ankle or tibial plafond injury on ipsilateral extremity
* BMI > 50
* Severe problems maintaining follow up
* Previous ankle/tibial plafond fracture
* Prisoners
* Neurological impairments that impair balance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Ankle Range of Motion (ROM) | 2 weeks after surgery
  maximum plantarflexion and maximum dorsiflexion
Ankle ROM | 6 weeks after surgery
  maximum plantarflexion and maximum dorsiflexion
Ankle ROM | 6 months after surgery
  maximum plantarflexion and maximum dorsiflexion

SECONDARY OUTCOMES:
Self reported subject compliance with exercise program: number of days completed | 2 weeks after surgery
  Comparison of compliance between a full American Academy of Orthopaedic Surgeons (AAOS) home exercise program/formal physical therapy visits and the simplified ankle dorsiflexion with a wooden block
Self reported subject compliance with exercise program: number of days completed | 6 weeks after surgery
  Comparison of compliance between a full AAOS home exercise program/formal physical therapy visits and the simplified ankle dorsiflexion with a wooden block
Lower Extremity Functional Scale score | 2 weeks after surgery.
  Comparison of Lower Extremity Functional Scale score (0 to 80 points) between and within groups. A higher score means better function.
Lower Extremity Functional Scale score | 6 weeks after surgery.
  Comparison of Lower Extremity Functional Scale score (0 to 80 points) between and within groups. A higher score means better function.
Lower Extremity Functional Scale score | 6 months after surgery.
  Comparison of Lower Extremity Functional Scale score (0 to 80 points) between and within groups. A higher score means better function.
Pain and ankle Range of Motion | 2 weeks after surgery
  Comparison of analog pain scores (Visual Analog Scale 0-100mm) between and within groups to gauge relationship of pain and ankle range of motion. Lower visual analog scale indicates less pain and higher Range of Motion means better ankle movement.
Pain and ankle Range of Motion | 6 weeks after surgery
  Comparison of analog pain scores (Visual Analog Scale 0-100mm) between and within groups to gauge relationship of pain and ankle range of motion. Lower visual analog scale indicates less pain and higher Range of Motion means better ankle movement.
Pain and ankle Range of Motion | 6 months after surgery.
  Comparison of analog pain scores (Visual Analog Scale 0-100mm) between and within groups to gauge relationship of pain and ankle range of motion. Lower visual analog scale indicates less pain and higher Range of Motion means better ankle movement.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Yarboro, MD, Principal Investigator — University of Virginia Orthopaedic Surgey
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No